CLINICAL TRIAL: NCT06405100
Title: Efficacy and Safety of Tacrolimus in Combination With Anti-CD20 Monoclonal Antibody (Ripertamab) in the Initial Treatment of Patients With Minimal Change Disease: a Multi-center Randomized Controlled Clinical Trial
Brief Title: Efficacy and Safety of Tacrolimus in Combination With Ripertamab in the Initial Treatment of Patients With MCD
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Collaborators: First Affiliated Hospital Xi'an Jiaotong University (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); The Second Affiliated Hospital of Air Force Military Medical University (Unknown); Shaanxi Provincial People's Hospital (Other); Shaanxi Provincial Hospital of Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Shiren sun, Chief, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAC and ripertamab in MCD
Record Dates: First submitted 2024-05-04; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Minimal Change Disease
MeSH Terms: conditions — Nephrosis, Lipoid | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): Supportive care+Prednisolone
  Interventions: Drug: Supportive care+Prednisone
- Test group 1 (Active Comparator): Supportive care+Tacrolimus+Ripertamab
  Interventions: Drug: Supportive care+Tacrolimus+Ripertamab
- Test group 2 (Active Comparator): Supportive care+Ripertamab
  Interventions: Drug: Supportive care+Ripertamab

INTERVENTIONS:
Drug: Supportive care+Prednisone — Supportive care: Control blood pressure:ACEI/ARB; Diet that is low in fat and salt; Stop smoking; Moderate exercise.
  Induction period: 1mg/kg/day. The maximum dose is not more than 60mg. The duration of adequate prednisone is a minimum of 4 weeks and a maximum of 16 weeks.
  Maintenance period: A reduction of 5-10mg/wk was initiated after 2 weeks of complete remission and finally discontinued after 6 months of maintenance at 5mg/day.
  Other Names: Control group
  Arms: Control Group
Drug: Supportive care+Tacrolimus+Ripertamab — Supportive care: Control blood pressure:ACEI/ARB; Diet that is low in fat and salt; Stop smoking; Moderate exercise.
  Tacrolimus：Induction period: 0.05mg/kg/d. It will be given in two doses 12 hours apart. The blood concentration should be up to 5-10ng/ml. Maintenance therapy was initiated two weeks after complete remission; Maintenance period: Reduced to a blood concentration of 3-8ng/ml, and stopped after 6 months of maintenance treatment.
  Ripertamab: Given twice every two weeks at a dose of 1000mg. 1000mg is added at 6 months.
  Other Names: Test group 1
  Arms: Test group 1
Drug: Supportive care+Ripertamab — Supportive care: Control blood pressure:ACEI/ARB; Diet that is low in fat and salt; Stop smoking; Moderate exercise.
  Ripertamab: Given twice every two weeks at a dose of 1000mg. 1000mg is added at 6 months.
  Other Names: Test group 2
  Arms: Test group 2

SUMMARY:
To evaluate the safety and efficacy of ripertamab and its combination with tacrolimus in the initial treatment of MCD to provide a treatment regimen with higher remission rates, lower recurrence rates, and fewer side effects in patients with MCD.

DETAILED DESCRIPTION:
Minimal change disease is the third most common primary kidney disease in adults with idiopathic nephrotic syndrome. The pathological features of the disease are no or only slight changes under light microscope, and the foot process fusion under electron microscope. The KDIGO guidelines recommend oral adequate doses of glucocorticoids as the initial treatment for adults with MCD. However, 48%-76% of patients relapse after tapering or gradual discontinuation of the drug, requiring a high cumulative dose of glucocorticoids. As the cumulative dose of glucocorticoids increases, the potential for side effects increases. In addition, 10% to 30% of patients frequently relapse, and 15% to 30% of these are steroid dependent. Therefore, the clinical goals for patients with MCD are to achieve early remission of proteinuria, reduce hormonal side effects, and more importantly, prevent the recurrence of proteinuria.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old;
2. Primary minimal change disease confirmed by renal biopsy (Initial therapy);
3. 24h-UTP>3.5g/d or PCR>3500mg/g, and serum albumin<30g/L;
4. Agree to participate in the project and sign the informed consent.

Exclusion Criteria:

1. Secondary minimal change disease;
2. eGFR<60 mL/min/1.73m2;
3. Had history of mental disease, dysnoesia, serious cardiovascular and cerebrovascular diseases, pulmonary insufficiency, malignant tumors or other major diseases that are not suitable for clinical experiments;
4. Active bleeding in the gastrointestinal tract;
5. Prior treatment with corticosteroids or other immunosuppressants;
6. HBV, HCV, HIV or other untreated infections, congenital or acquired immunodeficiency diseases;
7. Have been vaccinated with live vaccine in the past four weeks;
8. Serum bilirubin > 3.6mg/dl for at least 1 month or liver function ≥3 times the upper limit of normal value;
9. Allergic to prednisolone, tacrolimus, or ripertamab;
10. Reluctance to use contraception or plan pregnancy/lactation within 6 months of study completion;
11. Had history of alcohol/drug abuse;
12. Unable to give informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Relapse rate at 24 months | Up to 24 months after enrollment
  Relapse: Proteinuria>3.5g/d or PCR>3500mg/g after complete remission has been achieved.

SECONDARY OUTCOMES:
Relapse rate at 12/18 months | Up to 18 months after enrollment
  The relapse rates of MCD patients at 12 months and 18 months were observed
Partial or complete remission at 2/6/12/24 months | Up to 24 months after enrollment
  Partial remission: Reduction of proteinuria to 0.3-3.5g/d, or PCR 300-3500mg/g and a decrease >50% from baseline Complete remission: Reduction of proteinuria to <0.3g/d or PCR<300mg/g
The time from the start of treatment to achieve complete remission | Up to 24 months after enrollment
  The time it takes for patients with MCD to reach a state of complete remission needs to be observed
The time from clinical complete remission to replase | Up to 24 months after enrollment
Safety-adverse events | The time from randomization until the occurrence of such adverse events, up to 24 months
  Creatinine levels doubled from baseline; an increase ≥30% from eGFR baseline; ESRD; adverse events; drug-related adverse events, and abnormal clinical manifestations